CLINICAL TRIAL: NCT00879385
Title: Targeted Demethylation to Enhance Response or Overcome Resistance to EGFR Blocking Agents in KRAS Wild-type Metastatic Colorectal Cancer Patients Using Sequential Decitabine and Panitumumab
Brief Title: KRAS Wild-type Metastatic Colorectal Cancer Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Amgen (Industry); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI31116
Record Dates: First submitted 2009-04-08; First posted 2009-04-10 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Colorectal Cancer
Keywords: KRAS wild-type; Colon; Cancer; colorectal; metastatic colorectal; advanced colorectal
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — Decitabine; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Dacogen™ (decitabine); Drug: Vectibix® (panitumumab)

INTERVENTIONS:
Drug: Dacogen™ (decitabine) — Dacogen™ (decitabine) is a FDA approved drug (NDA - 021790) for the treatment of myelodysplastic syndromes (MDS) including previously treated and untreated, de novo and secondary MDS (refractory anemia, refractory anemia with ringed sideroblasts, refractory anemia with excess blasts, refractory anemia with excess blasts in transformation, and chronic myelomonocytic leukemia).
  Decitabine will be given on this study at 45 mg/m2 IV over 2 hrs
Drug: Vectibix® (panitumumab) — Vectibix® (panitumumab) is a FDA approved drug (BLA-125147) indicated as a single agent for the treatment of EGFR-expressing metastatic colorectal carcinoma with disease progression on or following fluoropyrimidine, oxaliplatin, and irinotecan chemotherapy regimens. Approval is based on progression-free survival; no data demonstrate an improvement in disease-related symptoms or increased survival.
  DRUG DESCRIPTION Vectibix® (panitumumab) is a recombinant, human IgG2 kappa monoclonal antibody that binds specifically to the human epidermal growth factor receptor (EGFR). Panitumumab has an approximate molecular weight of 147 kDa. Panitumumab is produced in genetically engineered mammalian (Chinese Hamster Ovary) cells.
  Panitumumab will be given on this study at 6 mg/kg, IV over 1 hr

SUMMARY:
OBJECTIVES:

Primary Objectives

1.To evaluate the safety and feasibility of the sequential use of a DNA methyltransferase (DNMT) inhibitor (decitabine) with a targeted biological agent against EGFR (panitumumab) for KRAS wild type tumors in the second or third line treatment of advanced metastatic colorectal cancer.

Secondary Objectives

1. To examine re-expression or a reduction in promoter methylation in genes involved in tumor suppressor pathways known to be important in colorectal cancer (CRC) or involved in EGFR signaling pathway.
2. Evaluate overall response (OR = CR +PR) according to RECIST criteria at 2, 4, and 6 cycles. Progression free survival, measured as the first evidence of tumor growth from the start of treatment will also be assessed.
3. Measure CEA levels at the beginning of each cycle to examine if they correlate with treatment response or disease progression.

DETAILED DESCRIPTION:
Patients with metastatic colorectal cancer are living longer and running out of therapeutic options due to disease resistance. Epidermal growth factor receptor (EGFR) has been validated as a therapeutic target in colorectal cancer (CRC). Ligand binding to EGFR activates the RAS/RAF/MAPK, STAT, and PI3K/AKT signaling pathways, which together modulate cellular proliferation, adhesion, migration, and survival. Anti-EGFR targeted antibodies cetuximab and panitumumab administered as monotherapy in CRC have shown response rates of approximately 9% and 17% respectively (Amado et al., 2008; Saltz et al., 2004). Single agent panitumumab has been approved for use in third line colorectal cancer and has been shown improve progression free survival over supportive care. Further subset analysis showed the response rate of 17% was confined to patients with KRAS wild type tumors only and that this group (approximately 60-70% of all CRC patients) should be considered for further study (Amado et al., 2008). According to the Huntsman Cancer Hospital registry, colorectal cancer patients are the largest disease group within our gastrointestinal cancer group and many have or eventually will progress on available therapy or are or will become intolerant to the side effects of second line therapies such as oxaliplatin neuropathy or irinotecan induced diarrhea, yet still are candidates for treatment.

In the lab through translational research studies, we hope to identify re-expression or a reduction in promoter methylation of genes involved in tumor suppressor pathways known to be important in colorectal cancer (CRC) or involved in EGFR signaling pathway. Candidate genes we will evaluate will include genes described in prior studies as associated with the CpG island methylator phenotype (CIMP) as well as genes previously reported to be hypermethylated in association with colorectal neoplasia. These will include APC, SFRP family members, CDH-1 (e-cadherin) and p16 (Belshaw et al., 2008; Lind et al., 2004; Suehiro et al., 2008). Other genes more specific to EGFR or KRAS signaling that will be assessed include: RASSF1A , a tumor suppressor gene know to be hypermethylated in several human cancers including CRC, is occasionally associated with KRAS wild type and when silenced by methylation allows for RAS activation (Kang et al., 2006; Oliveira et al., 2005); SOX17, a member of the transcription factor superfamily know to be hypermethylated in CRC and lead to disrupted Wnt signaling (Zhang et al., 2008); SOCS-1 a negative regulator of STAT3 an activating ligand for EGFR that has been shown to be silenced by hypermethylation and allow for constitutive signaling via EGFR (Lee et al., 2006); and PTEN, a tumor suppressor that antagonizes the PI3K- AKT/PKB signaling pathway by dephosphorylating phosphoinositides (Noro et al., 2007). Further candidate genes may be discovered or added based on preliminary data and ongoing research. Methylation analysis and gene expression pattern changes will be done using methylation specific PCR and bisulfite sequencing of genes known to be involved in EGFR signaling pathways and colorectal neoplasia as described above. We have prior data from our own work as well as others to suggest the use of a hypomethylating agent can resensitize colon cancer cells to therapeutic agents (Karpf et al., 1999; Morita et al., 2006). The translational component of this research will be supported by institutional translational grant awarded to the PI, Kimberly Jones, as of July 1st, 2008. This information may help identify other important targets and allow for the design of better combination therapies. We plan to do these assays on weekly blood and buccal samples while patients are on therapy, on epithelial cells swabbed from panitumumab associated skin rash, and on archived or biopsied tumor specimens when available (from KRAS testing (required) and optional end-of treatment biopsy).

The pharmacokinetic profile for decitabine has been well described and offers several possible dosing schedules feasible for clinical practice and combination with other agents. Decitabine is currently being tested in combination with standard cytotoxic agents. It has shown some activity in solid tumors, however, myelosuppression is a common side effect, especially when given concurrently with other myelosuppressive therapy (carboplatin) (Appleton et al., 2007; Plimack et al., 2007). We propose a novel study using decitabine in combination with a non-myelosuppressive targeted biological agent as well as giving it sequentially rather than concurrently to try to maximize the effect of the second drug by dosing it during the demethylation window. In the dose-finding study reported by Appleton et al., they recommended a dose of 90 mg/m2 over 6 hours every 28 days, but went up as high as 135 mg/m2 and combined this with carboplatin (Appleton et al., 2007). We have chosen a dose of 45 mg/m2 decitabine every 14 days based on its reported safety and biological equivalence from this study. There was no grade 3 or 4 hematological toxicities observed with 3 patients infused with 45 mg/m2 of decitabine followed by 5 AUC carboplatin; there was 1 episode of grade 3 leukopenia and 1 of grade 3 neutropenia in 4 patients infused with 45 mg/m2 of decitabine followed by 6 AUC carboplatin (Appleton et al., 2007). At the higher dose of 90 mg/m2 with 5 AUC carboplatin in 13 patients, 5 episodes of grade 4 leukopenia or neutropenia were observed; in 10 patients with 90 mg/m2 and 6 AUC carboplatin, there were 4 episodes of grade 4 leukopenia or neutropenia. The proposed infusion over 2 hours should not create any infusion rate toxicities and will be a schedule patients will tolerate. Daily lower dose infusions used in hematological disorders maybe be efficacious but daily intravenous chemotherapy impacts patient's quality of life significantly. Decitabine also has an elimination half-life of 30 minutes, so will clear the body rapidly. The proposed administration of the decitabine twice, at half the dose, in a 28-day period should be better tolerated than the 90 mg/m2 combined with carboplatin. The myelosuppressive toxicity which is the main toxicity of decitabine should be less significant as it is not being combined with a second myelosuppressive agent as it was with carboplatin. Low dose decitabine (45 mg/m2) has nearly equivalent hypomethylating effects to 90 mg/m2 in both blood and buccal cells. The more frequent dosing (every 2 weeks versus every 4 weeks) should maintain the hypomethylating effect at a lower dose. Additionally, we propose a novel dosing schedule where our second agent, panitumumab, will be given on alternating weeks and targeting the EGFR pathway when it is hypomethylated from the prior decitabine treatment. Our work as well as others, has demonstrated that specific promoter hypomethylation is observed by 8-14 days after the start of treatment and genomic DNA reverts to baseline levels by 28 to 35 days after the start of treatment (Appleton et al., 2007; Samlowski et al., 2005, Kantarjian, 2007 #23).

We will also be assessing clinical response and progression free survival (PFS) and comparing it to historical controls of patients treated with panitumumab monotherapy. If the combination can be given safely and responses are seen that are equal to or better than the single agent panitumumab data, we would plan a multi-center larger phase II trial.

ELIGIBILITY:
Inclusion Criteria:

1. At least third line stage IV metastatic colorectal cancer or metastatic colorectal cancer patients intolerant to second line therapy.
2. Tumor is KRAS wild-type.
3. ECOG performance status of 0-1
4. Age (≥)18
5. Adequate bone marrow function (ANC >1500/mm3, hemoglobin >9 g/dL (which may be obtained by transfusions or growth factor support), platelets >100,000)
6. Adequate hepatic function (AST and ALT <2.5x upper limit of normal (ULN), unless there are liver metastasis in which case AST and ALT <5.0 x ULN.
7. Adequate renal function (Serum creatinine ≤1.5 x ULN or calculated creatinine of >50 ml/min)
8. Timing of the last previous chemotherapy, radiotherapy, immunotherapy, and/or surgery treatment to be greater than 2 weeks before protocol entry
9. Patients are required to have recovered from side effects of prior treatment with the exception of neuropathy (to be determined by treating physician and NCI CTCAE grade <1)
10. Women of child-bearing age must be willing to use adequate contraception and have negative serum or urine pregnancy test within 3 days prior to registration.
11. Available archived tumor sample or provide consent for re-biopsy of tumor.
12. Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.
13. Patients must have at least one measurable site of disease according to RECIST criteria

Exclusion Criteria:

1. Prior treatment with decitabine.
2. Known hypersensitivity to decitabine and panitumumab or their excipients.
3. Any of the following within 6 months prior to drug administration: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, or cerebrovascular accident.
4. Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥2 that are independent of previous treatments.
5. Severely impaired lung function by medical history and/or clinical lung exam.
6. Any active (acute or chronic) or uncontrolled infection/ disorders.
7. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
8. Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
9. Hypertension that can not be controlled by medications (>170/100 mmHg)
10. Diagnosis of any secondary malignancy within the last 3 years (except basal cell carcinoma, squamous cell skin cancer, or stage I or less carcinoma fully treated)
11. Known HIV infection by patient disclosure or on active treatment.
12. Other severe acute or chronic medical or psychiatric condition or lab abnormality that would place the participant at excess risk by participating as judged by the study investigator.
13. Women of child-bearing age who are pregnant or lactating
14. History of noncompliance to medical regimens
15. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Evaluate safety & feasibility of sequential use of a DNA methyltransferase (DNMT) inhibitor (decitabine) with targeted biological agent against EGFR (panitumumab) for KRAS wild type tumors in second or third line treatment of colorectal cancer. | 2 years

SECONDARY OUTCOMES:
To examine re-expression or a reduction in promoter methylation in genes involved in tumor suppressor pathways known to be important in colorectal cancer (CRC) or involved in EGFR signaling pathway. | 2 years
Evaluate overall response (OR = CR +PR) according to RECIST criteria at 2, 4, and 6 cycles. Progression free survival, measured as the first evidence of tumor growth from the start of treatment will also be assessed. | 2 years
Measure CEA levels at the beginning of each cycle to examine if they correlate with treatment response or disease progression. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Sharma, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Garrido-Laguna I, McGregor KA, Wade M, Weis J, Gilcrease W, Burr L, Soldi R, Jakubowski L, Davidson C, Morrell G, Olpin JD, Boucher K, Jones D, Sharma S. A phase I/II study of decitabine in combination with panitumumab in patients with wild-type (wt) KRAS metastatic colorectal cancer. Invest New Drugs. 2013 Oct;31(5):1257-64. doi: 10.1007/s10637-013-9947-6. Epub 2013 Mar 17. PMID 23504398